CLINICAL TRIAL: NCT00524316
Title: A Phase II Study of SUNITINIB MALATE (Sutent) and Chemoembolization in Patients With Unresectable Hepatocellular Cancer
Brief Title: Sunitinib and Chemoembolization in Treating Patients With Liver Cancer That Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000563261; RPCI-I-82706
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-03

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Doxorubicin; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib (Experimental): oral sunitinib malate once daily on days 1-7 and 15-35 in course 1 and on days 1-28 in all subsequent courses
  Interventions: Drug: doxorubicin hydrochloride; Drug: sunitinib malate; Other: laboratory biomarker analysis; Procedure: hepatic artery embolization; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Transarterial chemoembolization
Drug: sunitinib malate — Given Orally
Other: laboratory biomarker analysis — Correlative Study
Procedure: hepatic artery embolization — Surgical procedure
Procedure: quality-of-life assessment — Correlative Study

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Chemoembolization kills tumor cells by blocking the blood flow to the tumor and keeping chemotherapy drugs, such as doxorubicin, near the tumor. Giving sunitinib together with chemoembolization may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving sunitinib together with chemoembolization works in treating patients with liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the progression-free survival at 4 months of patients treated with this regimen.

Secondary

* To determine overall survival of these patients.
* To determine if dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) can be used to measure decrease in tumor perfusion and vascular permeability as a result of treatment with sunitinib malate in combination with TACE, and if it can be useful in prognosis.
* To examine the safety and tolerability of this regimen.
* To determine if a change in circulating endothelial precursor cell number and total monocyte count on days 3, 8, 10, and 35 of therapy (as compared with levels at baseline) and decrease in soluble vascular endothelial growth factor receptor-2 in serum on days 8 (before TACE), 10, and 35 of therapy (as compared with baseline) correlate with improved response and survival.
* To determine the effect of this therapy on quality of life as measured by the FACT-HEP scale prior to each course of therapy.

OUTLINE: This is a multicenter study.

Patients receive oral sunitinib malate once daily on days 1-7 and 15-35 in course 1 and on days 1-28 in all subsequent courses. Patients undergo hepatic artery chemoembolization with doxorubicin hydrochloride on day 8 of course 1 only. Treatment with sunitinib malate repeats every 6 weeks* in the absence of disease progression or unacceptable toxicity.

NOTE: *Course 1 is 7 weeks in duration; all subsequent courses are 6 weeks in duration.

Blood samples are collected at baseline and periodically during study to measure circulating endothelial precursor cell levels, total monocyte count, and soluble vascular endothelial growth factor receptor-2.

Quality of life is assessed by the FACT-HEP scale at baseline, prior to each course of treatment, and then at the completion of treatment.

After completion of study treatment, patients are followed every 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically, cytologically, or serologically* confirmed hepatocellular carcinoma meeting the following criteria:

  * 1-4 lesions
  * Involvement of 1 or both liver lobes NOTE: *Alpha-fetoprotein (AFP) > 500 mcg/L in high-risk patients
* Measurable disease by CT scan or MRI

  * Disease does not exceed 50% of the liver parenchyma
  * At least 1 lesion ≥ 3 cm in longest diameter
* Tumor burden involves < 50% of the liver
* Refused surgery OR unresectable disease due to any of the following:

  * Multifocality
  * Advanced cirrhosis
  * Comorbid illness
* Candidate for chemoembolization
* No fibrolamellar histology
* No ascites
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Hemoglobin ≥ 8.5 g/dL (transfusion allowed)
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 2 mg/dL
* AST ≤ 5 times upper limit of normal (ULN)
* INR < 1.5
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 30 mL/min
* No bleeding diathesis or coagulopathy
* No active congestive heart failure
* No uncontrolled angina
* No myocardial infarction within the past 12 months
* No cardiac arrhythmia
* Ejection fraction ≥ 45% (in patients with known coronary artery disease and in patients > 50 years of age)
* Child-Pugh class A or B cirrhosis
* No impedance of hepatopedal blood flow (portal vein thrombosis)
* No thrombosis of the main portal vein
* No encephalopathy
* No biliary obstruction
* No variceal bleed within the past 6 months
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib malate
* No absolute contraindication to doxorubicin, iodinated contrast material, microfibrillar collage hemostat, or dexamethasone
* No other concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Psychiatric illness or social situation that would limit compliance with study requirements
* No other active malignancies within the past year except nonmelanoma skin cancer or carcinoma in situ
* No significant traumatic injury within the past 4 weeks
* No QTc prolongation (i.e., QTc interval ≥ 500 msec) or other significant ECG abnormalities
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after the completion of study treatment

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* Prior liver-directed therapy, such as chemoembolization, radiofrequency ablation, cryoablation, or ethanol injection allowed if the following criteria are met:

  * Treated lesion remains inactive by CT scan or MRI and new lesion being embolized is distinct from the previously treated lesion
  * Radiographic progression of previously treated lesion requiring re-embolization
* Prior liver resection allowed
* Prior immunotherapy allowed
* No prior antiangiogenesis therapy
* No prior liver transplantation

  * Patients awaiting a cadaveric or orthotopic liver transplantation are eligible provided they have end-stage liver disease with a priority score of < 20 points
* More than 4 weeks since prior radiotherapy or chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 4 weeks since prior major surgery or open biopsy
* At least 1 week since prior fine needle biopsy
* No concurrent immunotherapy
* No concurrent radiotherapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent therapeutic doses of coumarin-derivative anticoagulants (e.g., warfarin)

  * Doses of ≤ 1 mg/day are allowed for prophylaxis of thrombosis as long as INR ≤ 1.5
  * Both full dose and prophylactic dose low molecular weight heparin allowed as long as PT INR ≤ 1.5
* No anticipated major surgery during and for 3 months after completion of study treatment
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-04; Primary Completion 2010-12 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Iyer, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Sunitinib and Chemoembolization: Treatment: Cycle (C)1-Sunitinib 37.5mg po d1-7 followed by TACE with doxorubicin in lipodiol on d8, continued sunitinib 37.5mg po qd d15-36 followed by 2 weeks off. C2 onwards- sunitinib 4 weeks on and 2 weeks off, with dose escalation to 50 mg in pts without any grade 3 toxicities in C1.
Period: Overall Study
Arm/Group | Treatment: Sunitinib and Chemoembolization
Started | 16
Completed | 0
Not Completed | 16
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 7
Not completed — Disease Progression | 7

BASELINE CHARACTERISTICS:
Arm/Group | Treatment: Sunitinib and Chemoembolization
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: median progression free survival in months
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Population: All treated and eligible patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment: Sunitinib and Chemoembolization
Number analyzed (Participants) | 16
months | 8.0 [4.3 to 9.3]

2. Secondary Outcome: Overall Survival
Description: median survival in months
Time Frame: as for outcome 1
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment: Sunitinib and Chemoembolization
Number analyzed (Participants) | 16
months | 15.1 [6.3 to 24.5]

3. Secondary Outcome: Tissue Perfusion, Ktrans, IAUC, and Percent Viable Tumor as Measured by DCE-MRI at Baseline and on Days 8 (Before Transarterial Chemoembolization), 10, and 35
Time Frame: Baseline, day 8, day 10, day 28 and day 35
Population: Due to the study's early termination and inadequate number of patients, no data were collected for this Outcome Measure.
Arm/Group | Treatment: Sunitinib and Chemoembolization
Number analyzed (Participants) | 0

4. Secondary Outcome: Safety and Tolerability
Description: Number of participants with adverse advent.
  Please refer to adverse event reporting for more detail.
Time Frame: Daily while on treatment through study completion, an average of 1 year
Population: All treated and eligible patients
Measure: Number; unit: participants
Arm/Group | Treatment: Sunitinib and Chemoembolization
Number analyzed (Participants) | 16
participants | 16

5. Secondary Outcome: Assess the Change in the Quality of Life Among Patients Using the FACTHep (Version 4) for Hepatobiliary Cancers.
Description: We utilized the FACT-HEP TOTAL SCORE (version 4) quality-of-life scale, which is a 45 item scale ranging from 96-178. Higher scores reflect better quality of life.
  No subscales were analyzed.
Time Frame: Baseline and Cycle 2
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment: Sunitinib and Chemoembolization
Number analyzed (Participants) | 16
units on a scale
  Baseline | 143.6 (25.1)
  Cycle 2 | 136.8 (21.9)

6. Secondary Outcome: Tumor Marker Response (AFP)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Baseline, week 7 and every 6 weeks after
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment: Sunitinib and Chemoembolization
Number analyzed (Participants) | 16
percentage of participants | 13 [2 to 38]

ADVERSE EVENTS:
Arm/Group | Treatment: Sunitinib and Chemoembolization
Serious Adverse Events (participants affected / at risk) | 16/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Sunitinib and Chemoembolization (N=16)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (4)
Constipation (Gastrointestinal disorders) | 1 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (3)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Lipase increased (Investigations) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (3)
Confusional state (Psychiatric disorders) | 1 (3)
Renal failure (Renal and urinary disorders) | 1 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: Sunitinib and Chemoembolization (N=16)
Anaemia (Blood and lymphatic system disorders) | 11 (70)
Leukopenia (Blood and lymphatic system disorders) | 10 (82)
Lymphopenia (Blood and lymphatic system disorders) | 11 (127)
Neutropenia (Blood and lymphatic system disorders) | 7 (35)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (92)
Arrhythmia (Cardiac disorders) | 1 (3)
Tachycardia (Cardiac disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 2 (10)
Retinal haemorrhage (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (5)
Abdominal pain (Gastrointestinal disorders) | 13 (54)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (3)
Constipation (Gastrointestinal disorders) | 10 (34)
Diarrhoea (Gastrointestinal disorders) | 10 (41)
Dry mouth (Gastrointestinal disorders) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (5)
Dysphagia (Gastrointestinal disorders) | 2 (4)
Eructation (Gastrointestinal disorders) | 1 (3)
Flatulence (Gastrointestinal disorders) | 1 (3)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (5)
Gingival pain (Gastrointestinal disorders) | 1 (3)
Glossodynia (Gastrointestinal disorders) | 2 (4)
Lip dry (Gastrointestinal disorders) | 1 (3)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (51)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (6)
Stomatitis (Gastrointestinal disorders) | 5 (16)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (42)
Chills (General disorders) | 5 (13)
Cyst (General disorders) | 1 (1)
Fatigue (General disorders) | 15 (69)
Gait disturbance (General disorders) | 2 (4)
Influenza like illness (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 3 (5)
Oedema peripheral (General disorders) | 3 (3)
Pyrexia (General disorders) | 7 (23)
Cholangitis (Hepatobiliary disorders) | 1 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 8 (54)
Fungal infection (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 1 (6)
Infection (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (4)
Alanine aminotransferase increased (Investigations) | 9 (44)
Ammonia increased (Investigations) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 14 (107)
Blood alkaline phosphatase increased (Investigations) | 11 (46)
Blood amylase increased (Investigations) | 4 (25)
Blood bicarbonate decreased (Investigations) | 1 (3)
Blood bilirubin increased (Investigations) | 2 (9)
Blood creatinine increased (Investigations) | 4 (17)
Blood fibrinogen decreased (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 2 (6)
Lipase increased (Investigations) | 5 (24)
Weight decreased (Investigations) | 8 (20)
Anorexia (Metabolism and nutrition disorders) | 13 (56)
Dehydration (Metabolism and nutrition disorders) | 7 (21)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (16)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (28)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 (73)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (11)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 14 (71)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (27)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5)
Balance disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (15)
Drooling (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 6 (12)
Headache (Nervous system disorders) | 4 (10)
Leukoencephalopathy (Nervous system disorders) | 1 (3)
Neuropathy (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (11)
Syncope (Nervous system disorders) | 1 (3)
Anxiety (Psychiatric disorders) | 1 (3)
Confusional state (Psychiatric disorders) | 2 (4)
Depression (Psychiatric disorders) | 1 (3)
Hallucination, visual (Psychiatric disorders) | 1 (3)
Insomnia (Psychiatric disorders) | 3 (12)
Chromaturia (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Penis disorder (Reproductive system and breast disorders) | 1 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (19)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (5)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (5)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1 (2)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (9)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (3)
Hypertension (Vascular disorders) | 4 (6)
Hypotension (Vascular disorders) | 4 (12)
Orthostatic hypotension (Vascular disorders) | 1 (3)

LIMITATIONS AND CAVEATS:
Due to the study's early termination and inadequate number of patients, no patients were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes